CLINICAL TRIAL: NCT00814476
Title: The Efficacy, Short and Long Term Effects of Regular Home Use Vs Diabetic Team - Supported Use of the Medtronic CareLink Therapy Management System in Patients With Diabetes
Brief Title: The Effects of Regular Home Use Vs Diabetic Team- Supported Use of the Medtronic CareLink Therapy Management System.
Acronym: CareLink
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: rmc005047ctil
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Type 1 Diabetes
Keywords: Medtronic CareLink; therapy management; diabetes; insulin pump; Blood glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Regular treated group in the first segment and CareLink treated group in the second segment
  Interventions: Other: regular home use and Medtronic CareLink Therapy Management
- 1. CareLink team supported group (Experimental): CareLink team supported group
  Interventions: Other: Medtronic CareLink therapy management system

INTERVENTIONS:
Other: Medtronic CareLink therapy management system — At the first segment, the usage of the CareLink system will be accompanied by the diabetic team, through at least monthly contact via the internet initiated by the diabetic team. In the second phase of the study,during the following 4 months, there will be regular home use of the CareLink system, without support initiated by the diabetic team
  Arms: 1. CareLink team supported group
Other: regular home use and Medtronic CareLink Therapy Management — At the first 4 months patients will continue at their regular treatment and contacts initiated by the study team via internet/electronic mail will be made once a month. At the second segment of the study patients there will be home use of the CareLink System until the end of the study. No further contact will be initiated by the study team.
  Arms: 2

SUMMARY:
Randomized, two arms, controlled, open study comprised of two consecutive segments. At the first segment that will last during the first 4 months of the study, patients will be randomized to the Care link treated group or non Care link treated group. At this segment of the study the usage of the Care link system will be accompanied by the diabetic team, through at least monthly contact via the Internet initiated by the diabetic team. At the second segment of the study, during the following 4 months, both groups will use the Care link System, home-use, without support initiated by the diabetic team.

DETAILED DESCRIPTION:
A randomized, two arms, controlled, open study in order to compare the efficacy, short and long term effects of regular home-use Vs diabetic team- supported use of the Medtronic CareLink therapy management system in patients with diabetes.

Primary objective:

To assess the efficacy, short term (4 months) and long term (8 months) effects of using the Medtronic CareLink® Therapy Management System for Diabetes on the following parameters:

1. Metabolic control as expressed by HbA1c.
2. Hypoglycemic events- number and severity of episodes.
3. DKA and ketosis events- number and severity of episodes.
4. Patient's satisfaction and quality of life measured by treatment satisfaction and quality of life questionnaires.
5. 7 points glucose profile.

Secondary objective:

To compare the efficacy of 4 months treatment using the CareLink® Therapy Management System, accompanied with intensive contact (at least once a month) initiated by diabetic team via the internet/electronic mail Vs home use treatment - without monthly contact initiated by the diabetic team

Study design:

The study will be comprised of two consecutive segments. At the first segment that will last during the first 4 months of the study, patients will be randomized to the CareLink treated group or non CareLink treated group. At this segment of the study the usage of the CareLink system will be accompanied by the diabetic team, through at least monthly contact via the internet initiated by the diabetic team. At the second segment of the study, during the following 4 months, both groups will use the CareLink system, home-use, without support initiated by the diabetic team.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes diagnosed at least 6 months prior to study entry
2. Current treatment with Medtronic 722 /712 external insulin pump systems
3. Treatment with insulin pump at least 3 month prior to study entry
4. An internet access from patient's home
5. Age 0-35 years old
6. HbA1c>7.8
7. Signing inform consent forms

Exclusion Criteria:

1. Any significant disease or conditions, including psychiatric disorders that in the opinion of the investigator are likely to effect his compliance or ability to complete the study
2. Patients participating in other device or drug studies

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | At Baseline and every 4 month after

SECONDARY OUTCOMES:
Hypoglycemic events | will be recorded through the whole study period
DKA and ketosis events | will be recorded through the whole study period
Patient's satisfaction and quality of life questionnaire | At baseline visit and every 4 months after
7 points glucose profile | Will be recorded 2 days before baseline visit and every 4 months after

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Principal Investigator — Rabin Medical Center
Locations (1):
- Schnider children medical center, Petah Tikva, Israel